CLINICAL TRIAL: NCT06356636
Title: Impact of the Financial Inclusion Improves Sanitation and Health (FINISH) 2022- 2024 Intervention. Protocol for a Cluster - Randomized Controlled Trial in Kenya's Homa Bay County and Uganda's Kamwenge District
Brief Title: Impact of the Financial Inclusion Improves Sanitation and Health
Acronym: FINISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amref Health Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: P1216/2022
Record Dates: First submitted 2024-02-26; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: cluster; randomized controlled trial; sanitation; evaluation; open defecation; Uganda; Kenya
MeSH Terms: conditions — Behavior | interventions — Health

STUDY DESIGN:
Intervention Model Description: The participants are divided into two or more groups, with each group receiving a different intervention or a control condition. The outcomes of each group are compared at the end of the study to assess the effectiveness of the intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: to be updated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): The intervention arm involves communities within Homa Bay County in Kenya and Kamwenge District in Uganda, where the FINISH Mondial initiative is implemented. This intervention aims to improve sanitation and health through a public-private partnership model, engaging communities, governments, entrepreneurs, and financiers to enhance sanitation services and supply chains.
  Interventions: Behavioral: Financial Inclusion Improves Sanitation and Health
- Control group (No Intervention): The control arm includes communities in Siaya County in Kenya and Bushenyi in Uganda, where the FINISH intervention is not implemented, serving as a comparison to evaluate the effectiveness of the intervention.

INTERVENTIONS:
Behavioral: Financial Inclusion Improves Sanitation and Health — This innovative model engages transformative partnerships which include four key stakeholders (communities, communities, governments, entrepreneurs, and financiers) to improve sanitation services and supply value chains. The work is two-sided: to create demand for improved sanitation facilities in communities while facilitating microcredit access for people and sanitation businesses on the supply side.
  Arms: Treatment group

SUMMARY:
The goal of this interventional study is to evaluate the impacts of Financial Inclusion improvement sanitation and Health (FINISH) interventions in Kenya's Homa Bay County and Uganda's Kamwenge District among children under five. The main questions it aims to answer are:

1. What is the estimated impact of the FINISH model on health outcomes (diarrhoea occurrence and hygienic behaviour) as well as social (school attendance and sanitation) in the intervention groups?
2. What are the perspectives, attitudes, and practices of various stakeholders (communities, governments, entrepreneurs, and financiers) regarding the FINISH model?
3. What is the cost-effectiveness of the FINISH model, including the amount of leverage funds generated?

The FINISH model postulates that countries will be supported to improve the enabling business environment for sanitation, markets to offer improved safely managed services and products at an affordable price, and formal and informal financial institutions will offer more funding to businesses and households for satiation and hygiene.

Researchers will then compare intervention areas (Homa Bay in Kenya and Kamwenge in Uganda) with control areas (Siaya and Bushenyi in Kenya and Uganda, respectively) to see if the FINISH intervention leads to improved sanitation, health outcomes, and economic benefits.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the intervention study involve communities within specific geographic locations (Homa Bay County in Kenya and Kamwenge District in Uganda) targeted by the FINISH Mondial initiative.

Exclusion Criteria:

* to be updated

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study targets both males and females in the intervention sites
Enrollment: 1090 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health outcome, measured as, Proportion of households with diarrhoea occurrence in children under five years, and social outcome measured as proportion of households whose children missed school due to diarrhoea occurrence | 4 years, which includes baseline data collection, implementation and endline data collection
  Diarrhoea occurrence in children under 5 years is measured as:- In the past two weeks child/children under 5 years who have had three or more loose or watery stools. households whose children missed school due to diarrhoea occurrence, is measured as proportion of households whose children missed school due to diarrhoeal disease in the past 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Homa Bay county, Homa Bay, Kenya

IPD SHARING:
Plan to Share IPD: Yes